CLINICAL TRIAL: NCT00769925
Title: Improving Care for Anxiety in Pediatric Settings
Brief Title: Assessing Different Methods of Anxiety Care in Pediatric Settings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is transitioning to another institution
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K01MH072952 (NIH); K01MH072952 (NIH); DSIR 84-CTS
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Anxiety Disorders
Keywords: Generalized Anxiety; Social Phobia; Separation Anxiety; Phobia
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation; Phobic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapist Assisted Bibliotherapy-Primary Care (TAB-PC) (Experimental)
  Interventions: Behavioral: Therapist-Assisted Bibliotherapy-Primary Care
- Cognitive Behavior Therapy-Primary Care (CBT-PC) (Experimental)
  Interventions: Behavioral: Cognitive Behavior Therapy-Primary Care

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy-Primary Care — Children will receive cognitive behavioral therapy from a child anxiety specialist at their doctor's office (the primary care clinic). The children will learn skills to cope with fear and anxiety, and parents will learn how to support their children in using these new skills.
  Other Names: Cognitive-Behavioral Therapy; CBT; Family CBT
  Arms: Cognitive Behavior Therapy-Primary Care (CBT-PC)
Behavioral: Therapist-Assisted Bibliotherapy-Primary Care — Parents will receive educational workbooks and ongoing support over the phone from a child anxiety specialist to learn how to use cognitive behavioral therapy skills to manage their children's fears and worries.
  Other Names: Parent Training; Self-help; Therapist Assisted Bibliotherapy
  Arms: Therapist Assisted Bibliotherapy-Primary Care (TAB-PC)

SUMMARY:
This study will compare the effectiveness of delivering cognitive behavioral therapy for children with anxiety disorders through in-person contact versus through workbooks and telephone communication.

DETAILED DESCRIPTION:
Approximately 13% of adolescents aged 9 to 17 suffer from an anxiety disorder, which can cause disruptive fear, worry, or uneasiness that impairs their normal functioning. These anxiety disorders can include generalized anxiety disorder (GAD), phobias, panic disorder, and obsessive-compulsive disorder (OCD), and they often co-occur with a second anxiety disorder or another mental or behavioral disorder, like depression. Research on interventions such as cognitive behavioral therapy (CBT) indicates that these interventions are helpful to children who suffer from anxiety disorders, but are not always used. This study will examine the feasibility of implementing CBT for children between the ages of 8 and 13 in two different forms: through in-person contact at the pediatric primary care setting and through telephone-based contact.

Participants in this study will be randomly assigned to receive either cognitive behavioral therapy in primary care (CBT-PC) or therapist-assisted bibliotherapy in primary care (TAB-PC). In CBT-PC, participants will have therapy administered by a child anxiety specialist, and the parents of participants will learn how to support the new skills their children learn in therapy. In TAB-PC, parents will receive educational workbooks and ongoing support over the phone from a child anxiety specialist to learn how to use CBT skills to manage their children's fears and worries. Participation in this study will last 3 to 4 months, with therapy visits occuring once a week at the beginning and tapering to once every other week at the end of treatment. At pre-treatment, mid-treatment, post-treatment, and a 3-month follow-up, participants will undergo structured clinical interviews to assess their anxiety levels and the severity of their conditions.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for one of the following disorders: separation anxiety disorder, social phobia, generalized anxiety disorder, specific phobia, or obsessive-compulsive disorder
* Takes a medication and has maintained a stable dose for 3 months before baseline assessment
* Pediatric medical care is provided through one of the participating primary care clinics
* Parent and child are fluent in English

Exclusion Criteria:

* Presence of a life threatening condition or a medical illness that would make participation unsafe
* Diagnosed with bipolar disorder I, mental retardation, or autism or has psychotic symptoms
* Acutely suicidal or homicidal or exhibiting dangerous behavior
* Parents do not consent for diagnosis and progress to be shared with their child's primary care physician

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Clinical Severity Rating on Anxiety Diagnostic Interview Schedule for Children for primary anxiety disorder | Measured at pre-treatment and post-treatment

SECONDARY OUTCOMES:
Clinical Global Impression scale-Improvement Change | Measured at pre-treatment, mid-treatment, post-treatment, and a 3-month follow-up
Screening for Anxiety Related Emotional Disorders (SCARED) parent and child self-report scales | Measured at pre-treatment, mid-treatment, post-treatment, and a 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Chavira, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Chavira DA, Drahota A, Garland AF, Roesch S, Garcia M, Stein MB. Feasibility of two modes of treatment delivery for child anxiety in primary care. Behav Res Ther. 2014 Sep;60:60-6. doi: 10.1016/j.brat.2014.06.010. Epub 2014 Jul 11. PMID 25075802